CLINICAL TRIAL: NCT01807754
Title: Simulated Screening Study of Combined Digital X-Ray, Ultrasound and Photoacoustic Breast Imaging
Brief Title: Simulated Screening Study for Breast Imaging
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul L. Carson Ph.D, Principal Investigator, University of Michigan
Other Study IDs: HUM 00069294; 2R01CA091713 (NIH)
Record Dates: First submitted 2012-12-06; First posted 2013-03-08 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Breast Cysts; Breast Tumors
Keywords: automated ultrasound imaging (AUS); digital breast tomosynthesis (DBT); photoacoustic imaging (PAT)
MeSH Terms: conditions — Breast Cyst; Breast Neoplasms | interventions — X-Rays; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imaging scans for breast cancer screening: To simulate the performance of the combination of three new breast imaging systems to digital mammography and hand-held ultrasound that are currently used to find and evaluate breast masses.
  These three different systems make images of the breast in several ways to find breast masses and to distinguish normal and abnormal masses. This may result in less unnecessary call-backs from mammography.
  Interventions: Procedure: X-ray and ultrasound imaging scanning; Procedure: Photoacoustic imaging scans for breast cancer screening

INTERVENTIONS:
Procedure: X-ray and ultrasound imaging scanning — Digital tomosynthesis mammogram uses a low radiation dose, taking x-ray pictures of the breast from many angles to make a 3D(dimensional)image. The participant will be seated and her breast positioned as in a normal mammogram, though with reduced pressure. The x-ray tube will move quickly above the breast to take the images. Then, an ultrasound scan will be done using gel on your breast to assist in acquiring quality imaging.
  Other Names: Digital tomosynthesis mammogram and automated ultrasound
Procedure: Photoacoustic imaging scans for breast cancer screening — The participant will be seated in front of the laser device with the breast positioned on the laser device platform. Each subject will be given a laser protective eye mask/goggles to wear and will be instructed how to wear the mask/goggles during the scan. In addition pulse monitor leads may be placed on the participant's chest to allow the computer to record ultrasound blood flow in the breast. The low intensity laser light will be focused on the targeted area of the breast.
  Other Names: Optoacoustic Imaging

SUMMARY:
This is a pilot, simulated breast cancer screening study. The goal of the study is to explore these scanning modalities:

1) Combined digital breast tomosynthesis(DBT)/dual-sides 3 dimensional-automated ultrasound(AUS)

2. Explore the utility of photoacoustic imaging as an adjunct to digital breast tomosynthesis(DBT)/ultrasound(US)alone.

DETAILED DESCRIPTION:
This is a pilot, simulated breast cancer screening study. In a population enriched with mammographic call-backs, we will study whether:

1) Combined digital breast tomosynthesis(DBT)/dual-sides 3 dimensional-automated ultrasound(AUS)will result in a lower call-back rate than digital breast tomosynthesis(DBT)alone.

2. Explore the utility of photoacoustic imaging as an adjunct to digital breast tomosynthesis(DBT)/ultrasound(US)alone.

This study will compare two new breast imaging systems to digital mammography and hand-held ultrasound that are commonly used to find and evaluate breast masses. Images will be done with digital breast tomosynthesis (DBT) and 3-D automated ultrasound(AUS) which will be done in the breast imaging clinic of the main hospital followed by the second light and ultrasound imaging that will be completed in the research lab.

ELIGIBILITY:
Inclusion Criteria:

* Women with possible masses
* All women should have had mammograms at University of Michigan Health System within 1 year before this research study.

Exclusion Criteria:

* Women who are physically unable to tolerate the length of the scan.
* Women who are less than 30 years of age or older than 80 years of age
* Women who are pregnant or lactating
* Women whose mass is in an area of the breast which makes it difficult to see in the research scans
* Womens with a single diagnosis of mammographic calcifications
* Women who have had a breast cancer with lumpectomy
* Women who are prisoners
* Women who are students or staff of investigators
* Women who cannot give consent
* Women with mammograms classified as probably benign because of follow-up of a recent benign biopsy.
* Women with breast pain who have been categorized as BIRADS(Breast Imaging Reporting and Data System) category 0(incomplete) on their most recent mammograms.
* Males, because their breast tissue is not easily imaged and numbers of potential cases are too few.

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population includes women who have had a mammogram at University of Michigan within one year who have been referred to the study. Participants may have a breast mass, either benign or cancerous.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-12; Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of new breast imaging devices | 3 years
  To determine if photoacoustic imaging is an adjunct to standard of care imaging with regards to quality of imaging. and ultrasound modalities and to determine if combining digital breast tomosynthesis and 3 dimensional automated ultrasound will result in a lower call-back ratio than imaging with digital breast tomosynthesis alone.

SECONDARY OUTCOMES:
Determining the ratio of "patient call backs" | 5 years
  To determine if combining digital breast tomosynthesis and 3 dimensional automated ultrasound will result in a lower call-back ratio than imaging with digital breast tomosynthesis alone.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L Carson, PhD, Principal Investigator — Univ. of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No